CLINICAL TRIAL: NCT02119104
Title: Prevenar (13v) Infant Drug Use Investigation (Regulatory Post Marketing Commitment Plan)
Brief Title: Prevenar (13v) Infant Drug Use Investigation
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1851122
Record Dates: First submitted 2014-03-05; First posted 2014-04-21 (Estimated); Results first posted 2017-06-19 (Actual); Last update posted 2017-06-19 (Actual); Status verified 2017-03

CONDITIONS: Infants
MeSH Terms: interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prevenar (13v)
  Interventions: Drug: Prevenar (13v)

INTERVENTIONS:
Drug: Prevenar (13v) — Prevenar (13v)

SUMMARY:
The purpose of this study is to investigate post marketing use and safety of Prevnar ( 13v) in infants vaccinated for the first time at the age of 2 months, inclusive, to 7 months, exclusive.

DETAILED DESCRIPTION:
The investigation will be conducted using the continuous investigation method, with which a satisfying registration conditions will be continuously registered until the number of contracted cases is reached.

ELIGIBILITY:
Inclusion Criteria:

* Vaccinees who meet all of the following conditions at the time of the first vaccination among infants who use Prevenar 13 in accordance with the indication, and dosage and administration of the vaccine will be included in the investigation:
* Infants aged 2 months, inclusive, to 7 months, exclusive
* Infants with no history of administration of pneumococcal vaccines including Prevenar 13
* Infants expected to receive 4 vaccinations

Exclusion Criteria:

* Vaccines must not be performed if the vaccinee corresponds to any of the following:
* Persons in whom a past history of anaphylaxis due to an ingredient of Prevenar 13 or diphtheria toxoid is evident
* Persons with evident pyrexia
* Persons who evidently have serious acute diseases
* Besides the persons listed above, persons who are in a status inappropriate for immunization

Ages: 2 Months to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Vaccinees who meet all of the following conditions at the time of the first vaccination among infants who use Prevenar 13 in accordance with the indication, and dosage and administration of the vaccine will be included in the investigation.
Sampling Method: Probability Sample
Enrollment: 1087 (Actual)
Dates: Start 2014-03; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1851122&StudyName=Prevenar%20%2813v%29%20Infant%20Drug%20Use%20Investigation

RESULTS

PARTICIPANT FLOW:
Groups:
- Prevenar 13: Participants were vaccinated with Prevenar 13 as follows: for primary immunization, three doses of Prevenar 13 0.5 mL were injected subcutaneously with an interval of at least 27 days between each dose. For booster immunization, one dose of Prevenar 0.5 mL was injected subcutaneously, at least 60 days after the third dose.
Period: Overall Study
Arm/Group | Prevenar 13
Started | 1087
Completed | 1071
Not Completed | 16
Not completed — Protocol Violation | 16

BASELINE CHARACTERISTICS:
Population: In total, 1087 participants were registered in this study. Of the 1087 participants, 16 participants were excluded from the safety analysis for the reasons of protocol violation.
Arm/Group | Prevenar 13
Number analyzed (Participants) | 1071
Age, Customized [Number; unit: Participants] — at the time of the first vaccination
  Participants
    2 to less than 3 months | 937
    3 to less than 4 months | 106
    4 to less than 5 months | 21
    5 to less than 6 months | 4
    6 to less than 7 months | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 501
  Male | 570

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Reactions
Description: An adverse reaction (vaccine-related adverse event) was any untoward medical occurrence which was considered to be related to Prevenar 13 in a participant who received Prevenar 13.
Time Frame: The entire observation period was from Day 1 of the 1st vaccination through Day 28 of the 4th vaccination.
Population: The safety analysis population comprised of participants who had received Prevenar 13 at least once and provided the safety data and who did not meet the exclusion criteria for the safety analysis.
Measure: Number; unit: Participants
Arm/Group | Prevenar 13
Number analyzed (Participants) | 1071
Participants
  Adverse Reactions | 432
  Serious Adverse Reactions | 3

ADVERSE EVENTS:
Description: The frequency of adverse events. The same event may appear as both an adverse event and a serious adverse event. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Prevenar 13
Serious Adverse Events (participants affected / at risk) | 11/1071
Other Adverse Events (participants affected / at risk) | 1026/1071
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prevenar 13 (N=1071)
Adenovirus infection (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 1
Respiratory syncytial virus bronchitis (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 1
Febrile convulsion (Nervous system disorders) | 1
Seizure (Nervous system disorders) | 1
Kawasaki's disease (Vascular disorders) | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1.0% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prevenar 13 (N=1071)
Somnolence (Nervous system disorders) | 36
Mood altered (Psychiatric disorders) | 47
Pyrexia (General disorders) | 248
Vaccination site erythema (General disorders) | 283
Vaccination site swelling (General disorders) | 248
Pharyngitis (Infections and infestations) | 13
Bronchitis (Infections and infestations) | 16
Insomnia (Psychiatric disorders) | 11
Irritability (Psychiatric disorders) | 12
Asthma (Respiratory, thoracic and mediastinal disorders) | 14
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 29
Diarrhoea (Gastrointestinal disorders) | 14
Eczema (Skin and subcutaneous tissue disorders) | 20
Erythema (Skin and subcutaneous tissue disorders) | 13
Vaccination site pain (General disorders) | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.